CLINICAL TRIAL: NCT01551979
Title: Therapeutic Efficacy of Cerebellar Repetitive Transcranial Magnetic Stimulation in Patients With Schizophrenia
Brief Title: Therapeutic Efficacy of Transcranial Magnetic Stimulation in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Sidney R. Baer, Jr. Foundation (Other)
Responsible Party: Principal Investigator, Mark Halko, Instructor in Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011P000373
Record Dates: First submitted 2012-03-01; First posted 2012-03-13 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; repetitive Transcranial Magnetic Stimulation
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active rTMS (Active Comparator): High frequency rTMS stimulation of the vermis(lobule VII) of the cerebellum.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Sham rTMS (Sham Comparator): Sham rTMS to the vermis (lobule VII) of the cerebellum.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — intermittent Theta Burst (iTBS) pattern (20 trains of 10 bursts given with 8s intervals) will be applied at 80% of active motor threshold. Each participant will receive 600 pulses per session.
  Sham participants will undergo the same procedures as those in the active rTMS group.
  Other Names: Transcranial Magnetic Stimulation; Noninvasive Brain Stimulation

SUMMARY:
The aim of this study is to look at the effectiveness of repetitive transcranial magnetic stimulation (rTMS) as a therapeutic intervention for patients with schizophrenia. The primary outcome is improvement in negative symptoms related to schizophrenia. The investigators are focusing on negative symptoms given their greater resistance to pharmacological and other established therapies. If the investigators trial were to show beneficial effects, its clinical significance would be great.

DETAILED DESCRIPTION:
This study builds on the results of a previous phase 1, single-site study in which we demonstrated the safety of image-guided theta burst stimulation (TBS) form of rTMS over the cerebellar vermis (Demirtas-Tatlidede et al., 2010) in eigh patients with schizophrenia.

The primary goal of the present study is to assess efficacy of iTBS to the cerebellar vermis on positive and negative symptoms of schizophrenia. A second, added goal is to investigate the mechanisms of the expected clinical improvement.

Schizophrenia is a leading cause of mental disability and current treatments still remain only partially successful for many patients. Our underlying hypothesis is that modulation of the cerebellar vermis may enhance activity of the neural systems that sub-serve cognition and emotion, reestablish the disturbed cerebellar regulation in schizophrenic patients, and produce clinical improvement.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years
* Diagnosis of schizophrenia according to DSM-IV criteria (Diagnostic and Statistical Manual) by a board-certified psychiatrist

Exclusion Criteria:

* Preexisting or progressive neurological disorders
* Prior neurological procedures
* Previous head injury
* Change in antipsychotic medication during the last 4 weeks
* Been an inpatient in a psychiatry clinic within the last month
* Any other axis 1 diagnosis
* Patients may not be actively enrolled in a separate intervention study
* Patients unable to undergo a brain MRI
* Any unstable medical condition
* History of seizures, diagnosis of epilepsy, history of abnormal (epileptiform_ EEG, or family history of treatment resistant epilepsy
* Possible pregnancy. All female participants of child bearing age are required to have a pregnancy test.
* Any metal in the brain, skull, or elsewhere unless approved by the responsible MD
* Any medical devices (ie. cardiac pacemaker, deep brain stimulator, medication infusion pump, cochlear implant, vagal nerve stimulator) unless otherwise approved by the responsible MD
* Substance abuse (alcohol, amphetamines, cocaine, MDMA [methylenedioxymethamphetamine], ecstasy, PCP [phencyclidine], Angle dust) or dependence within the past six months
* No medication is an absolute exclusion from TMS. Medications will be reviewed by the responsible MD and a decision about inclusion will be made based on the following: the patient's past medical history, drug dose, history of recent medication changes or duration of treatment, and combination with other CNS (central nervous system) active drugs (the published TMS guidelines review of medications to be considered with TMS)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Halko, Ph.D., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Batini C, Buisseret-Delmas C, Corvisier J, Hardy O, Jassik-Gerschenfeld D. Brain stem nuclei giving fibers to lobules VI and VII of the cerebellar vermis. Brain Res. 1978 Sep 22;153(2):241-61. doi: 10.1016/0006-8993(78)90405-5. PMID 80249
- [Background] Demirtas-Tatlidede A, Freitas C, Cromer JR, Safar L, Ongur D, Stone WS, Seidman LJ, Schmahmann JD, Pascual-Leone A. Safety and proof of principle study of cerebellar vermal theta burst stimulation in refractory schizophrenia. Schizophr Res. 2010 Dec;124(1-3):91-100. doi: 10.1016/j.schres.2010.08.015. PMID 20817483
- [Background] Demirtas-Tatlidede A, Freitas C, Pascual-Leone A, Schmahmann JD. Modulatory effects of theta burst stimulation on cerebellar nonsomatic functions. Cerebellum. 2011 Sep;10(3):495-503. doi: 10.1007/s12311-010-0230-5. PMID 21132574
- [Background] Fregni F, Boggio PS, Valle AC, Rocha RR, Duarte J, Ferreira MJ, Wagner T, Fecteau S, Rigonatti SP, Riberto M, Freedman SD, Pascual-Leone A. A sham-controlled trial of a 5-day course of repetitive transcranial magnetic stimulation of the unaffected hemisphere in stroke patients. Stroke. 2006 Aug;37(8):2115-22. doi: 10.1161/01.STR.0000231390.58967.6b. Epub 2006 Jun 29. PMID 16809569
- [Background] Fregni F, Thome-Souza S, Bermpohl F, Marcolin MA, Herzog A, Pascual-Leone A, Valente KD. Antiepileptic effects of repetitive transcranial magnetic stimulation in patients with cortical malformations: an EEG and clinical study. Stereotact Funct Neurosurg. 2005;83(2-3):57-62. doi: 10.1159/000086674. Epub 2005 Jun 30. PMID 15990468
- [Background] Fregni F, Freedman S, Pascual-Leone A. Recent advances in the treatment of chronic pain with non-invasive brain stimulation techniques. Lancet Neurol. 2007 Feb;6(2):188-91. doi: 10.1016/S1474-4422(07)70032-7. PMID 17239806
- [Background] George MS, Wassermann EM, Williams WA, Callahan A, Ketter TA, Basser P, Hallett M, Post RM. Daily repetitive transcranial magnetic stimulation (rTMS) improves mood in depression. Neuroreport. 1995 Oct 2;6(14):1853-6. doi: 10.1097/00001756-199510020-00008. PMID 8547583
- [Background] George MS, Nahas Z, Kozel FA, Goldman J, Molloy M, Oliver N. Improvement of depression following transcranial magnetic stimulation. Curr Psychiatry Rep. 1999 Dec;1(2):114-24. doi: 10.1007/s11920-999-0020-2. PMID 11122913
- [Background] Gershon AA, Dannon PN, Grunhaus L. Transcranial magnetic stimulation in the treatment of depression. Am J Psychiatry. 2003 May;160(5):835-45. doi: 10.1176/appi.ajp.160.5.835. PMID 12727683
- [Background] Hajak G, Marienhagen J, Langguth B, Werner S, Binder H, Eichhammer P. High-frequency repetitive transcranial magnetic stimulation in schizophrenia: a combined treatment and neuroimaging study. Psychol Med. 2004 Oct;34(7):1157-63. doi: 10.1017/s0033291704002338. PMID 15697042
- [Background] Hashimoto M, Ohtsuka K. Transcranial magnetic stimulation over the posterior cerebellum during visually guided saccades in man. Brain. 1995 Oct;118 ( Pt 5):1185-93. doi: 10.1093/brain/118.5.1185. PMID 7496779
- [Background] Heath RG. Modulation of emotion with a brain pacemamer. Treatment for intractable psychiatric illness. J Nerv Ment Dis. 1977 Nov;165(5):300-17. PMID 303280
- [Background] Heath RG, Dempesy CW, Fontana CJ, Myers WA. Cerebellar stimulation: effects on septal region, hippocampus, and amygdala of cats and rats. Biol Psychiatry. 1978 Oct;13(5):501-29. PMID 728506
- [Background] Huber TJ, Schneider U, Rollnik J. Gender differences in the effect of repetitive transcranial magnetic stimulation in schizophrenia. Psychiatry Res. 2003 Aug 30;120(1):103-5. doi: 10.1016/s0165-1781(03)00170-7. PMID 14500119
- [Background] Jardri R, Lucas B, Delevoye-Turrell Y, Delmaire C, Delion P, Thomas P, Goeb JL. An 11-year-old boy with drug-resistant schizophrenia treated with temporo-parietal rTMS. Mol Psychiatry. 2007 Apr;12(4):320. doi: 10.1038/sj.mp.4001968. No abstract available. PMID 17389898
- [Background] Jin Y, Potkin SG, Kemp AS, Huerta ST, Alva G, Thai TM, Carreon D, Bunney WE Jr. Therapeutic effects of individualized alpha frequency transcranial magnetic stimulation (alphaTMS) on the negative symptoms of schizophrenia. Schizophr Bull. 2006 Jul;32(3):556-61. doi: 10.1093/schbul/sbj020. Epub 2005 Oct 27. PMID 16254067
- [Background] Martin PI, Naeser MA, Theoret H, Tormos JM, Nicholas M, Kurland J, Fregni F, Seekins H, Doron K, Pascual-Leone A. Transcranial magnetic stimulation as a complementary treatment for aphasia. Semin Speech Lang. 2004 May;25(2):181-91. doi: 10.1055/s-2004-825654. PMID 15118944
- [Background] Ohtsuka K, Enoki T. Transcranial magnetic stimulation over the posterior cerebellum during smooth pursuit eye movements in man. Brain. 1998 Mar;121 ( Pt 3):429-35. doi: 10.1093/brain/121.3.429. PMID 9549519
- [Background] Papez JW. A proposed mechanism of emotion. 1937. J Neuropsychiatry Clin Neurosci. 1995 Winter;7(1):103-12. doi: 10.1176/jnp.7.1.103. No abstract available. PMID 7711480
- [Background] Pascual-Leone A, Rubio B, Pallardo F, Catala MD. Rapid-rate transcranial magnetic stimulation of left dorsolateral prefrontal cortex in drug-resistant depression. Lancet. 1996 Jul 27;348(9022):233-7. doi: 10.1016/s0140-6736(96)01219-6. PMID 8684201
- [Background] Rollnik JD, Huber TJ, Mogk H, Siggelkow S, Kropp S, Dengler R, Emrich HM, Schneider U. High frequency repetitive transcranial magnetic stimulation (rTMS) of the dorsolateral prefrontal cortex in schizophrenic patients. Neuroreport. 2000 Dec 18;11(18):4013-5. doi: 10.1097/00001756-200012180-00022. PMID 11192620
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Schmahmann JD. The role of the cerebellum in cognition and emotion: personal reflections since 1982 on the dysmetria of thought hypothesis, and its historical evolution from theory to therapy. Neuropsychol Rev. 2010 Sep;20(3):236-60. doi: 10.1007/s11065-010-9142-x. Epub 2010 Sep 7. PMID 20821056
- [Background] Schutter DJ, van Honk J, d'Alfonso AA, Peper JS, Panksepp J. High frequency repetitive transcranial magnetic over the medial cerebellum induces a shift in the prefrontal electroencephalography gamma spectrum: a pilot study in humans. Neurosci Lett. 2003 Jan 16;336(2):73-6. doi: 10.1016/s0304-3940(02)01077-7. PMID 12499043
- See also: Related Information — http://tmslab.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 22 patients gave informed consent for the study during the initial screening visit. After patients were found ineligible to participate following review of medical records, withdrew consent, or were lost to follow-up, only 17 remained for the randomization phase and started the study.
Groups:
- Active rTMS: High frequency rTMS stimulation of the vermis(lobule VII) of the cerebellum.
  Repetitive Transcranial Magnetic Stimulation: intermittent Theta Burst (iTBS) pattern (20 trains of 10 bursts given with 8s intervals) will be applied at 80% of active motor threshold. Each participant will receive 600 pulses per session.
  Sham participants will undergo the same procedures as those in the active rTMS group.
- Sham rTMS: Sham rTMS to the vermis (lobule VII) of the cerebellum.
  Repetitive Transcranial Magnetic Stimulation: intermittent Theta Burst (iTBS) pattern (20 trains of 10 bursts given with 8s intervals) will be applied at 80% of active motor threshold. Each participant will receive 600 pulses per session.
  Sham participants will undergo the same procedures as those in the active rTMS group.
Period: Overall Study
Arm/Group | Active rTMS | Sham rTMS
Started | 10 | 7
Last Day of Treatment (After 5 Days) | 10 | 7
1 Week Post Treatment | 10 | 6
Completed | 8 | 5
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active rTMS | Sham rTMS | Total
Number analyzed (Participants) | 10 | 7 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 7 | 17
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 8 | 5 | 13
Region of Enrollment [Number; unit: participants]
  United States | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on the Positive and Negative Syndrome Scale (PANSS) Positive Subscale
Description: Therapeutic efficacy was evaluated with the Positive and Negative Syndrome Scale (PANSS) Positive Subscale, a 7 item subscale measuring the presence/absence and severity of positive symptoms of schizophrenia. The minimum score is 7 and the maximum score is 49, with higher values representing greater symptom severity. Change from baseline on the PANSS Positive Subscale can range from -42 to +42; negative values represent an improvement in symptom severity, and positive values represent worsening symptom severity. Therapeutic efficacy was assessed at baseline, after 5 days of treatment, 1 week post treatment, and 3 weeks post treatment.
Time Frame: Before treatment (baseline), last day of treatment (after 5 days of treatment), 1 and 3 weeks post treatment
Population: Participant drop out
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 10 | 7
units on a scale
  5 days of treatment - baseline | -2.4 (3.565) | -1.857 (1.574)
  1 week post treatment - baseline: number analyzed (Participants) | 9 | 6
  1 week post treatment - baseline | -5.889 (3.333) | -3.667 (3.724)
  3 week post treatment - baseline: number analyzed (Participants) | 8 | 5
  3 week post treatment - baseline | -5 (4.504) | -3 (3.317)

2. Primary Outcome: Change From Baseline on the Positive and Negative Syndrome Scale (PANSS) Negative Subscale
Description: Therapeutic efficacy was evaluated with the Positive and Negative Syndrome Scale (PANSS) Negative Subscale, a 7 item subscale measuring the presence/absence and severity of negative symptoms of schizophrenia. The minimum score is 7 and the maximum score is 49, with higher values representing greater symptom severity. Change from baseline on the PANSS Negative Subscale can range from -42 to +42; negative values represent an improvement in symptom severity, and positive values represent worsening symptom severity. Therapeutic efficacy was assessed at baseline, after 5 days of treatment, 1 week post treatment, and 3 weeks post treatment.
Time Frame: Before treatment (baseline), last day of treatment (after 5 days of treatment), 1 and 3 weeks post treatment
Population: Participant drop out
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 10 | 7
units on a scale
  5 days of treatment - baseline | -1 (4.876) | -1.571 (2.070)
  1 week post treatment - baseline: number analyzed (Participants) | 9 | 6
  1 week post treatment - baseline | -3.889 (3.296) | -1.667 (3.141)
  3 week post treatment - baseline: number analyzed (Participants) | 8 | 5
  3 week post treatment - baseline | -3.5 (6.024) | -0.2 (4.604)

3. Primary Outcome: Change From Baseline on the Positive and Negative Syndrome Scale (PANSS) General Subscale
Description: Therapeutic efficacy was evaluated with the Positive and Negative Syndrome Scale (PANSS) General Subscale, a 16 item subscale measuring the presence/absence and severity of general psychopathology of schizophrenia. The minimum score is 16 and the maximum score is 112, with higher values representing greater psychopathology severity. Change from baseline on the PANSS General Subscale can range from -96 to +96; negative values represent an improvement in symptom severity, and positive values represent worsening symptom severity. Therapeutic efficacy was assessed at baseline, after 5 days of treatment, 1 week post treatment, and 3 weeks post treatment.
Time Frame: Before treatment (baseline), last day of treatment (after 5 days of treatment), 1 and 3 weeks post treatment
Population: Participant drop out
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 10 | 7
units on a scale
  5 days of treatment - baseline | -3.1 (4.149) | -2.714 (5.090)
  1 week post treatment - baseline: number analyzed (Participants) | 9 | 6
  1 week post treatment - baseline | -8.222 (5.696) | -2 (4.690)
  3 week post treatment - baseline: number analyzed (Participants) | 8 | 5
  3 week post treatment - baseline | -7.375 (10.127) | 0 (1)

4. Primary Outcome: Change From Baseline on the Clinical Global Impression (CGI) Severity of Illness
Description: Treatment response was evaluated with the Clinical Global Impressions (CGI) Scale, which is comprised of two companion one-item measures that use 7-point scales to evaluate severity of psychopathology and improvement from the initiation of treatment; each component is rated separately and the CGI does not yield a global score. The CGI Severity of Illness is a 7-point subscale in which a clinician rates the severity of the patient's illness at the time of assessment. Ratings range from 1 to 7 and higher values represent more severe psychopathology: 1 indicates a normal and not at all ill patient and 7 indicates among the most extremely ill patients. Change from baseline on the CGI Severity of Illness subscale can range from -6 to +6, with negative values representing an improvement in psychopathology and positive values representing worsening psychopathology. Severity of Illness was assessed at baseline, after 5 days of treatment, 1 week post treatment, and 3 weeks post treatment.
Time Frame: Before treatment (baseline), last day of treatment (after 5 days of treatment), 1 and 3 weeks post treatment
Population: Participant drop out
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 10 | 7
units on a scale
  5 days of treatment - baseline | -0.3 (0.483) | -0.286 (0.488)
  1 week post treatment - baseline: number analyzed (Participants) | 10 | 6
  1 week post treatment - baseline | -0.4 (0.699) | -0.5 (0.548)
  3 week post treatment - baseline: number analyzed (Participants) | 8 | 5
  3 week post treatment - baseline | -0.5 (0.535) | -0.2 (0.837)

5. Primary Outcome: Clinical Global Impression (CGI) Global Improvement
Description: Treatment response was evaluated with the Clinical Global Impressions (CGI) Scale, which is comprised of two companion one-item measures that use 7-point scales to evaluate severity of psychopathology and improvement from the initiation of treatment; each component is rated separately and the CGI does not yield a global score. The CGI Global Improvement is a 7-point subscale in which a clinician assesses how much a patient's illness has changed compared to baseline. Ratings range from 1 to 7, with 1 indicating very much improved and 7 indicating very much worse. Change from baseline on the CGI Global Improvement subscale can range from -6 to +6, with negative values representing an improvement in psychopathology and positive values representing worsening psychopathology. Global Improvement was assessed after 5 days of treatment, 1 week post treatment, and 3 weeks post treatment.
Time Frame: Last day of treatment (after 5 days of treatment), 1 and 3 weeks post treatment
Population: Participant drop out
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 10 | 7
units on a scale
  5 days of treatment | 3.6 (0.516) | 3.429 (1.134)
  1 week post treatment: number analyzed (Participants) | 10 | 6
  1 week post treatment | 3.3 (0.675) | 4 (0.632)
  3 week post treatment: number analyzed (Participants) | 8 | 5
  3 week post treatment | 3.375 (0.518) | 3.8 (0.447)

6. Secondary Outcome: Change From Baseline on the Calgary Depression Scale for Schizophrenia
Description: The Calgary Depression Scale for Schizophrenia is a 9-item scale that assesses depressive symptoms in patients with schizophrenia. Each item is rated separately and ratings range from 0 to 3. Higher values represent more severe depressive symptoms: 0 indicates an absent symptom and 3 indicates a severe symptom. The overall Calgary Depression Scale score is computed by summing each item. The total Calgary Depression Scale score ranges from 0 to 27, with higher values representing more severe depression in patients with schizophrenia. Change from baseline on the Calgary Depression Scale can range from -27 to +27, with negative values representing an improvement in depressive symptoms and positive values representing worsening depressive symptom severity. Depression was assessed at baseline, after 5 days of treatment, 1 week post treatment, and 3 weeks post treatment.
Time Frame: Before treatment (baseline), last day of treatment (after 5 days of treatment), 1 and 3 weeks post treatment
Population: Participant drop out
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 10 | 7
units on a scale
  5 days of treatment - baseline: number analyzed (Participants) | 10 | 6
  5 days of treatment - baseline | -2.6 (3.204) | -1.167 (2.563)
  1 week post treatment - baseline: number analyzed (Participants) | 10 | 6
  1 week post treatment - baseline | -2.7 (2.908) | -1.833 (2.229)
  3 week post treatment - baseline: number analyzed (Participants) | 8 | 5
  3 week post treatment - baseline | -2.25 (2.121) | 0.8 (2.387)

ADVERSE EVENTS:
Time Frame: 4 weeks (5 days of treatment and 1 week and 3 weeks post treatment)
Description: 0 total number of participants at risk for all-cause mortality because all-cause mortality was not collected/assessed.
Arm/Group | Active rTMS | Sham rTMS
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/7
Other Adverse Events (participants affected / at risk) | 5/10 | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active rTMS (N=10) | Sham rTMS (N=7)
Acute exacerbation of psychosis (Psychiatric disorders) | 1 (1) | 0 (0) — Acute exacerbation of psychosis was assessed to be possibly related to participation in the study, but likely not related to the TMS. Subject was hospitalized.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active rTMS (N=10) | Sham rTMS (N=7)
Discomfort with TMS (Nervous system disorders) | 1 (1) | 0 (0) — Discomfort with the TMS-EEG measures being done at baseline in the frontal lobe area. Discomfort was assessed to be related to the study.
Blood pressure increase (Cardiac disorders) | 1 (1) | 0 (0) — Blood pressure elevation was assessed to be possibly related to the study.
Headache (Nervous system disorders) | 2 (2) | 1 (2) — Headaches were reported during EEG measures during baseline assessment, pre-TMS, and post-TMS. Headaches were assessed as possibly or probably related to the study.
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) — Scalp pain reported as pressure on scalp over the ears and top of head. Scalp pain was assessed as possibly related to the study.
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) — Neck pain reported due to dystonia or heaviness of the coil. Neck pain due to dystonia was assessed as not related to study participation. Neck pain due to the coil was assessed as probably related to the study.
Head heaviness (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) — Heaviness was reported on right side of head during and after TMS. Headache was assessed to be possibly related to the study.
Change in energy level (Nervous system disorders) | 1 (2) | 0 (0) — Subject reported being mildly or moderately tired post-TMS.
Change in mood (Psychiatric disorders) | 1 (1) | 0 (0) — Subject reported feeling depressed. Change in mood assessed to be possibly related to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No